CLINICAL TRIAL: NCT07259031
Title: Postoperative Effects of Phrenic Nerve Paralysis Induced During Resection Surgery: A Prospective Study With Electromyography
Brief Title: Postoperative Effects of Intraoperative Temporary Phrenic Nerve Paralysis in Lung Resection Surgery
Acronym: PNCrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ferdane Melike Duran (Other)
Responsible Party: Sponsor-Investigator, Ferdane Melike Duran, Assistant professor of Thoracic Surgery, Konya City Hospital
Organization: Konya City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU2019-1421; NEU2019-1421 (Other: Necmettin Erbakan University Faculty of Medicine Ethics Commitee)
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Prolonged Air Leak; Phrenic Nerve; EMG
Keywords: residual air space; prolonged air leak; Phrenic nerve crush; Diaphragm electromyography

STUDY DESIGN:
Intervention Model Description: This study was designed as a parallel, two-arm interventional trial comparing patients undergoing lobectomy with or without brief intraoperative phrenic nerve compression. Participants were assigned to either the experimental group (phrenic nerve compression for 1-2 seconds) or the control group (no phrenic nerve manipulation). Postoperative respiratory function, diaphragmatic EMG findings, and clinical follow-up parameters were compared between the groups.
Masking Description: This is an open-label study. Participants, surgeons, and outcome assessors are aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phrenic crush (Experimental): Patients underwent standard lobectomy via muscle-sparing thoracotomy with brief intraoperative compression (1-2 seconds) of the phrenic nerve to induce transient diaphragmatic paralysis.
  Interventions: Procedure: İntraoperative phrenic nerve compression
- Control (No Intervention): Patients underwent standard lobectomy via muscle-sparing thoracotomy without any intraoperative manipulation or compression of the phrenic nerve.

INTERVENTIONS:
Procedure: İntraoperative phrenic nerve compression — Temporary intraoperative compression (1-2 seconds) of the phrenic nerve during lobectomy to induce transient diaphragmatic paralysis and minimize postoperative residual space.
  Arms: Phrenic crush

SUMMARY:
This prospective clinical study aimed to evaluate the postoperative effects of temporary phrenic nerve paralysis induced by intraoperative phrenic nerve crush during lung resection surgery. The study compared postoperative pulmonary function, diaphragm activity, and clinical outcomes between patients who underwent intraoperative phrenic nerve crush and those who did not. The objective was to assess the reversibility, safety, and clinical impact of temporary phrenic nerve paralysis in relation to postoperative residual pleural space and prolonged air leak.

DETAILED DESCRIPTION:
This prospective observational study was conducted at the University of Health Sciences, Konya City Hospital, Department of Thoracic Surgery, between September 2019 and March 2023. The study included patients who underwent lung resection surgery via muscle-sparing thoracotomy. In the intervention group, a controlled intraoperative phrenic nerve crush was applied to induce temporary phrenic nerve paralysis. In the control group, no phrenic nerve manipulation was performed.

The primary objective was to evaluate the postoperative effects and reversibility of temporary phrenic nerve paralysis using diaphragm electromyography (EMG) and pulmonary function tests (FEV1, FVC). Secondary objectives included the assessment of residual pleural space filling, prolonged air leak, chest tube duration, and length of hospital stay. The study also aimed to determine whether temporary phrenic nerve paralysis could help minimize postoperative residual pleural space and prolonged air leak without causing permanent functional impairment.

Ethical approval for the study was obtained from the Necmettin Erbakan University Faculty of Medicine Ethics Committee (approval number: NEU2019-1421). Written informed consent was obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+) who underwent lobectomy via muscle sparing thoracotomy

  * Patients with adequate preoperative pulmonary function to tolerate lobectomy
  * Patients who provided written informed consent for participation.
  * Patients with available postoperative follow-up data, including EMG and pulmonary function tests

Exclusion Criteria:

* Patients who underwent wedge resection, segmentectomy, pneumonectomy, or VATS procedures
* Patients with previous phrenic nerve injury, diaphragmatic paralysis, or neuromuscular disorders affecting respiratory muscles.
* Patients with incomplete postoperative follow-up or missing EMG/PFT data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic Electromyography | Preoperative; 3 weeks postoperative; 6 months postoperative
  Quantitative assesment of diaphragmatic muscle activity using preoperative and postoperative EMG, recorded as motor unit action potential amplitude (mA) and duration (ms), to evaluate the degree of diaphragmatic dysfunction or recovery following intraoperative phrenic nerve compression.
Pulmonary Function Test - FEV1 | Preoperative; 3 weeks postoperative; 6 months postoperative
  Spirometric assessment of forced expiratory volume in 1 second (FEV1) to evaluate postoperative respiratory performance and the potential impact of brief intraoperative phrenic nerve compression. FEV1 values will be recorded as absolute volume (L) and as percent predicted (% predicted). Comparisons will be made between groups at each time point.
Pulmonary Function Test - FVC | Preoperative; 3 weeks postoperative; 6 months postoperative
  Spirometric assessment of forced vital capacity (FVC) to evaluate postoperative respiratory performance and the potential impact of brief intraoperative phrenic nerve compression. FVC values will be recorded as absolute volume (L) and as percent predicted (% predicted). Comparisons will be made between groups at each time point.

SECONDARY OUTCOMES:
Chest Tube Duration | Up to postoperative day 30
  Duration of chest tube placement recorded as the number of postoperative days from the time of insertion until removal. Comparisons will be made between groups.
Length of Hospital Stay | Up to postoperative day 30
  Total duration of hospitalization recorded as the number of days from the day of surgery until discharge. Comparisons will be made between groups.
Prolonged Air Leak | Up to postoperative day 30
  Incidence of prolonged postoperative air leak, defined as an air leak lasting more than 5 days after surgery. The outcome will be recorded as the number of participants with and without prolonged air leak in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdane M Duran, MD, Principal Investigator — University of Health Science, Konya City Hospital
Locations (1):
- Konya City Hospital, Department of Thoracic Surgery, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
İndividual participant data will not be shared because the study includes patient-specific clinical and electrophysiological data that cannot be fully anonymized. Data will only be used for the analysis described in the approved protocol.